CLINICAL TRIAL: NCT05499949
Title: The Franciscus Obesity NASH Study
Acronym: FONS
Status: Active, not recruiting | Type: Observational
Sponsor: Franciscus Gasthuis (Other)
Collaborators: Amsterdam UMC (Other); Erasmus Medical Center (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: FONS
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: NAFLD; NASH - Nonalcoholic Steatohepatitis; Obesity, Morbid
Keywords: Transient elastography; Bariatric surgery
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood Feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FONS group: Patients with morbid obesity enrolled for bariatric surgery in the Franciscus Gasthuis, Rotterdam, the Netherland
  Interventions: Diagnostic Test: NASH screening; Diagnostic Test: Cardiac dysfunction screening; Diagnostic Test: Liver biopsy

INTERVENTIONS:
Diagnostic Test: NASH screening — Evaluate liver steatosis and elasticity using transient elastography in the FONS group
Diagnostic Test: Cardiac dysfunction screening — Evaluate cardiac dysfunction in 60 patients from the FONS group with transthoracic echocardiography
Diagnostic Test: Liver biopsy — For participants from the FONS group with an elevated liver fibrosis measurement (≥F2) with TE, a laparoscopic liver biopsy will be performed during the bariatric procedure.

SUMMARY:
The purpose of this study is to evaluate Non-Alcoholic Fatty Liver Disease (NAFLD) and Non-Alcoholic Steatohepatitis (NASH) changes in terms of steatosis and elasticity in patients with morbid obesity 1, 3 and 5 years after bariatric surgery.

In addition, genomics, microbiome and metabolomics analyses will be carried out.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, 300 eligible patients will be included.

All participants will undergo lifestyle intervention before bariatric surgery. Extensive cardiometabolic analyses will be carried out. At 5 different moments (twice before and 3 times after bariatric surgery), liver steatosis and elasticity will be evaluate using Fibroscan. For those with an elevated liver fibrosis measurement (TE ≥7.2 kilopascal with M probe or ≥7.95 kilopascal with extra large probe), a laparoscopic liver biopsy will be performed during surgery. Patients will undergo gastric sleeve resection, Roux-n-Y gastric bypass or gastric minibypass.

ELIGIBILITY:
Inclusion Criteria:

Participants must fulfil all of the inclusion criteria (unless otherwise specified) for enrolment in the study.

1. Participants must fulfil the criteria of the International Federation for the Surgery of Obesity (IFSO) at screening.
2. Participants must be able to understand the nature of the study and written informed consent must be obtained before any study specific interventions are performed.

The cardiac function of a subset group of 30 subjects aged 35 years and older with low transient elastography measurements (≤F1) and no known cardiac disease, hypertension or diabetes mellitus will be compared with a similar number of patients with high transient elastography measurements (≥F3) and no known cardiac disease, hypertension or diabetes mellitus. These patients will be consecutively included.

The investigators will perform a liver biopsy during endoscopic bariatric surgery in the patients with an elevated transient elastography measurement (≥F2; suggesting fibrosis and therefore the presence of NASH) in order to correlate the histological diagnosis to the clinical diagnosis based on elastography. In those patients in whom the diagnosis of NASH is confirmed by histology, more detailed follow up in a separate program at the department of gastroenterology is indicated according to the current guidelines.

Exclusion Criteria:

Patients who meet any of the following criteria at screening (unless otherwise specified) will be excluded from the study:

1. Participants younger than 18 years or older than 65 years
2. Participants with an established diagnosis of liver pathology like, but not limited to:

   1. Hepatitis B
   2. Hepatitis C
   3. Autoimmune hepatitis
   4. Wilson's disease
   5. Hemochromatosis
   6. Primary biliary cholangitis
   7. Primary sclerosing cholangitis
   8. Alcoholic liver disease
3. Histologically documented liver cirrhosis (fibrosis stage F4), at screening or in a historical biopsy.
4. Participants with active HIV infection and/or treatment.
5. Participants with diagnosed malignancies with or without active treatment.
6. Participants with a history or evidence of any other clinically significant condition or planned or expected procedure that in the opinion of the investigator, may compromise the patient's safety or ability to complete the study.
7. The participant does not understand Dutch.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with morbid obesity enrolled for bariatric surgery at the Franciscus Gasthuis, Rotterdam, the Netherlands.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in liver steatosis (in decibel/meter) 5 years after bariatric surgery | baseline (enrolment) and 5 years after bariatric surgery
  Transient elastography is a non invasive test evaluating liver steatosis
Change from baseline in liver fibrosis (in kilopascal) 5 years after bariatric surgery | baseline (enrolment) and 5 years after bariatric surgery
  Transient elastography is a non invasive test evaluating liver fibrosis

SECONDARY OUTCOMES:
Change from baseline in liver steatosis (in decibel/meter) after lifestyle intervention | baseline (enrolment) and 3 months later
  Transient elastography is a non invasive test evaluating liver steatosis
Change from baseline in liver fibrosis (in kilopascal) after lifestyle intervention | baseline (enrolment) and 3 months later
  Transient elastography is a non invasive test evaluating liver fibrosis
Change from baseline in liver steatosis (in decibel/meter) 1 year after bariatric surgery | baseline (enrolment) and 1 year after bariatric surgery
  Transient elastography is a non invasive test evaluating liver steatosis
Change from baseline in liver fibrosis (in kilopascal) 1 year after bariatric surgery | baseline (enrolment) and 1 year after bariatric surgery
  Transient elastography is a non invasive test evaluating liver fibrosis
Change from baseline in liver steatosis (in decibel/meter) 3 years after bariatric surgery | baseline (enrolment) and 3 years after bariatric surgery
  Transient elastography is a non invasive test evaluating liver steatosis
Change from baseline in liver fibrosis (in kilopascal) 3 years after bariatric surgery | baseline (enrolment) and 3 years after bariatric surgery
  Transient elastography is a non invasive test evaluating liver fibrosis
Change from baseline in liver steatosis (in decibel/meter) according to the type of bariatric surgery | baseline and 1 and 3 years after bariatric surgery
  To evaluate if the type of bariatric surgery (gastric sleeve resection, Roux-en-Y Gastric bypass, Gastric minibypass) influences the steatosis in patients with morbid obesity, measured 1 and 3 years after bariatric surgery, adjusted for baseline steatosis/elasticity.
Change from baseline in liver fibrosis (in kilopascal) according to the type of bariatric surgery | baseline and 1 and 3 years after bariatric surgery
  To evaluate if the type of bariatric surgery (gastric sleeve resection, Roux-en-Y Gastric bypass, Gastric minibypass) influences the elasticity in patients with morbid obesity, measured 1 and 3 years after bariatric surgery, adjusted for baseline steatosis/elasticity.
Change from baseline in liver steatosis (in decibel/meter) according to the genetic profile | baseline and 1 year after surgery
  To determine if candidate genetic markers (PNPLA3, TM6SF2, MBOAT7, GCKR and HSD17B13) are associated to changes in NAFLD/NASH severity in patients with morbid obesity one year after bariatric surgery.
Change from baseline in liver fibrosis (in kilopascal) according to the genetic profile | baseline and 1 year after surgery
  To determine if candidate genetic markers (PNPLA3, TM6SF2, MBOAT7, GCKR and HSD17B13) are associated to changes in NAFLD/NASH severity in patients with morbid obesity one year after bariatric surgery.
Change from baseline in liver steatosis (in decibel/meter) according to gender and ethnicities | baseline and 1, 3 and 5 years after bariatric surgery
  To determine if liver steatosis differs between gender or ethnicities before bariatric surgery and the changes 1, 3 and 5 years after bariatric surgery
Change from baseline in liver fibrosis (in kilopascal) according to gender and ethnicities | baseline and 1, 3 and 5 years after bariatric surgery
  To determine if liver elasticity differs between gender or ethnicities before bariatric surgery and the changes 1, 3 and 5 years after bariatric surgery
Change from baseline in liver steatosis liver steatosis (in decibel/meter) according to the gut microbiota | baseline and 1 year after bariatric surgery
  To investigate the change in the ratio of Firmicutes/Bacteroides in the distal gut microbiota in patients with morbid obesity with NAFLD/NASH 1 year after bariatric surgery and the effects of these changes on transient elastography measurements.
Change from baseline in liver steatosis liver fibrosis (in kilopascal) according to the gut microbiota | baseline and 1 year after bariatric surgery
  To investigate the change in the ratio of Firmicutes/Bacteroides in the distal gut microbiota in patients with morbid obesity with NAFLD/NASH 1 year after bariatric surgery and the effects of these changes on transient elastography measurements.
Association between NAFLD/NASH and vascular dysfunction | baseline
  To determine if the presence of NAFLD/NASH before bariatric surgery is associated with (subclinical) vascular dysfunction using the carotid intima media thickness and pulse wave velocity
Association between NAFLD/NASH and cardiac dysfunction | baseline and 1 year after bariatric surgery
  To determine if the presence of NAFLD/NASH before bariatric surgery is associated with (subclinical) cardiac dysfunction using transthoracic echocardiography
Association between change in NAFLD/NASH and change in cardiac dysfunction | baseline and 1 year after bariatric surgery
  To determine if change of liver fibrosis stage is associated to change in cardiac function 1 year after bariatric surgery
Correlation between histology and transient elastography measurement in a population with morbid obesity | during surgery
  To establish the correlation between histology (liver biopsy) and transient elastography measurement in a population with morbid obesity

CONTACTS AND LOCATIONS:
Locations (1):
- Franciscus Gasthuis, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data are available upon reasonable request. The data that will be shared is individual participant data that underlie the results reported in the study, after deidentification (text, tables, figures and appendices). Also, the study protocol will be available. Data will be available beginning 9 months and ending 36 months following publication, for researchers who provide a methodologically sound proposal for any purpose. Proposals may be directed to w.theel@franciscus. nl up to 36 months following article publication. After 36 months, the data will be available in our hospital's data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Derived] Theel WB, Boxma-de Klerk BM, Dirksmeier-Harinck F, van Rossum EF, Kanhai DA, Apers JA, van Dalen BM, De Knegt RJ, Neecke B, van der Zwan EM, Grobbee DE, Hankemeier T, Wiebolt J, Castro Cabezas M. Effect of bariatric surgery on NAFLD/NASH: a single-centre observational prospective cohort study. BMJ Open. 2023 Jul 3;13(7):e070431. doi: 10.1136/bmjopen-2022-070431. PMID 37400234